CLINICAL TRIAL: NCT02412410
Title: Optimizing Sleep/Wake Related Cognitive Efficacy in Laborist Shifts: Toward Establishing Models of Safer Obstetrical Care
Brief Title: Optimizing Sleep/Wake Related Cognitive Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Margaret L. Dow, M.D., Assistant Professor Obstestrics-Gynecology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-008496
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Laborist; Sleep; Cognition; Fatigue
Keywords: laborist; efficacy; sleep; fatigue; SAFTE; cognition
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): Single arm pilot study analyzing sleep data and calculated efficacy before and after fatigue avoidance education (comparator is same group after intervention)
  Interventions: Behavioral: Fatigue avoidance education

INTERVENTIONS:
Behavioral: Fatigue avoidance education — Grand Rounds presentation of consequences of fatigue and fatigue avoidance techniques

SUMMARY:
This is a pilot study designed to elucidate sleep/wake patterns and associated cognitive efficacy of laborists involved in shift work at Mayo Clinic Rochester.

DETAILED DESCRIPTION:
Each of the ten physicians working laborist shifts will be asked to wear an actigraphy watch (ReadiBand- Fatigue Science, Vancouver, BC) continually for three weeks in the winter 2014-2015 for initial data collection. A brief sleep education intervention based on aerospace and military fatigue countermeasure training will be given at a one hour departmental grand rounds presentation on April 20, 2015. This intervention will be based on ACGME requirements for fatigue education for residents and will also address the latest data on sleep and health, as well as fatigue countermeasures of nap recommendations, sleep banking, and sleep hygiene. An additional two weeks of data will then be collected.

Data will be de-identified and entered into the Fatigue Science algorithm, which is validated to detect sleep quantity and quality. This algorithm allows labelling of data to reflect which type of shift, as well as its sequence in the schedule. For example, sleep/wake cycles of the fourth night shift of a series can be identified as such, so that wakefulness during a fourth night shift is not artificially compared to wakefulness during a first night of night shifts. Average efficacy during each type of shift, as well as average efficacy during each shift in a series of one type of shift can then be calculated. Efficacy is reported as a percentage, based on a nomogram established through military wakefulness task exercises and validated to correlate with blood alcohol level and with likelihood of human factor accident risk through the Department of Defense, US Army, US Navy, US Marine Corps, and Federal Railroad Association.

Calculated data on shift efficacy will significantly contribute to the growing literature on the strengths of the laborist model, and will help with internal schedule structure to continue to maximize efficacy. As laborist programs develop and expand, the investigators may also be forerunners in describing optimal scheduling and staffing for programs of similar size and scope. Ultimately, additional studies will use this innovative technology to elucidate the assumed but not scientifically established relationship between sleep/wake based cognitive efficacy and patient safety by superimposing the investigators' wakefulness data on the investigators' tracked adverse events. This would be landmark in the investigators' field and has the potential to effect groundbreaking safety measures in the investigators' training and staffing.

ELIGIBILITY:
Physicians working in Laborist role, exclusion only by subject declining participation

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Optimizing efficacy through fatigue avoidance -Comparison of calculated efficacy scores before and after fatigue avoidance education | 3 months
  Comparison of calculated efficacy scores before and after fatigue avoidance education

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Dow, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No